CLINICAL TRIAL: NCT02847234
Title: Factors Associated With Complications of Cervical Necrotizing Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0500
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Necrotizing Fasciitis
Keywords: Cervical necrotizing fasciitis; mediastinitis
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cervical necrotizing fasciitis (CNF) is a rare but severe complication of pharyngeal or dental infections. The infection can rapidly descend into the mediastinum and lead to a life-threatening prognosis. Treatment consists of a multidisciplinary approach in intensive care with radiologist and with early and repeated surgical debridement. Anti-inflammatory drugs have been incriminated by authors in the development of necrotizing fasciitis. Recently, a single-center study demonstrated that pharyngeal source of CNF and oral glucocorticoid intake before admission was associated with the occurrence of mediastinitis.

The aim of the study is to assess the incidence and factors associated with CNF complications, in particular mediastinitis. Secondary outcome is to describe patient characteristics, medical and surgical management.

Methods: A retrospective, observational, non-interventional multicentre study is conducted in nine intensive care units in France from January 2005 to December 2016.

ELIGIBILITY:
Inclusion Criteria:

- Patient admitted in ICU for management of cervical necrotizing fasciitis between 2005 and 2016.

Exclusion Criteria:

* Patients admitted in ICU for management of cervical abscess without cervical necrotizing fasciitis
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in ICU for management of cervical necrotizing fasciitis
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
incidence of mediastinitis | At the entry in ICU (Day 1)
  Computed tomography (CT) is performed at admission. Mediastinitis is described on CT finding.

SECONDARY OUTCOMES:
factors associated with mediastinitis | At the entry in ICU (Day 1)
  Computed tomography (CT) is performed at admission. Mediastinitis is described on CT finding.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rimmelé, MD PhD, Principal Investigator — Intensive Care unit, Edouard Herriot Hospital, 69003 Lyon, FRANCE
Locations (1):
- Intensive Care unit, Edouard Herriot Hospital, Lyon, France